CLINICAL TRIAL: NCT06080282
Title: Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology
Brief Title: Role of the Kallikrein-kinin System in Septic Cardiomyopathy
Status: Recruiting | Type: Observational
Sponsor: Qin Zhang (Other)
Responsible Party: Sponsor-Investigator, Qin Zhang, phd, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB202308109
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Sepsis
Keywords: sepsis; Septic cardiomyopathy; KKS
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples Without DNA — Excess blood from patient blood gas analysis, followed by separation of plasma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sepsis: No intervention

SUMMARY:
The purpose of this study is to investigate whether there are differential expressions of molecules in the kallikrein-kinin system (KKS) pathway in septic cardiomyopathy, and to analyze their regulatory mechanisms and gene expression changes.

DETAILED DESCRIPTION:
This study is designed as a prospective, single-center, prospective case-control study. The research plan mainly aims to collect clinical data and blood samples from patients with septic cardiomyopathy and the control group within the next 3 years (October 2023 to October 2025). Diagnostic criteria are as follows: (1) Diagnosis of sepsis is based on the SEPSIS 3.0 criteria, which is defined as a rapid increase in SOFA score by ≥2 points after infection as a clinical criterion for sepsis-related organ dysfunction. (2) Diagnostic criteria for septic cardiomyopathy include: diagnosis of sepsis and elevation of cardiac markers [cardiac troponin I (cTnI) or BNP]; systolic dysfunction: echocardiography shows LVEF < 50%; diastolic dysfunction: Doppler ultrasound shows an E/A ratio (rapid filling phase/atrial contraction phase) ≤1 at the mitral valve; BNP > 200 pg/mL; left ventricular fractional shortening (FS) > 25%; normal or increased wall thickness, decreased left ventricular filling rate.

ELIGIBILITY:
Inclusion Criteria:

(1) Age range greater than 18 years. (2) Patients diagnosed with septic cardiomyopathy. (3) Clear determination of the cause of myocardial injury, such as the source of infection, bacterial culture results, etc. (4) Patients who are capable of cooperating and completing the necessary examinations and treatments.

-

Exclusion Criteria:

(1) Presence of other significant underlying cardiovascular diseases, such as coronary heart disease, heart failure, etc. (2) Presence of other organ dysfunction that poses a significant threat to life, such as respiratory failure, liver failure, etc. (3) Presence of severe infections or inflammatory diseases unrelated to myocardial injury, such as severe acute pancreatitis. (4) History of receiving interventional treatments, such as immunomodulatory agents, anti-inflammatory drugs, etc. (5) Pregnant or lactating women. (6) Pediatric patients who are under the age of majority.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis and patients diagnosed with septic cardiomyopathy.
Sampling Method: Probability Sample
Enrollment: 640 (Estimated)
Dates: Start 2014-10-01 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2025-10-14 (Estimated)

PRIMARY OUTCOMES:
Survival | 28 days
  Survival

SECONDARY OUTCOMES:
Cardiac function | 24 hour
  Echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: QIN Zhang, phd, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China